CLINICAL TRIAL: NCT02977299
Title: Augmentation Versus Switch: Comparative Effectiveness Research Trial for Antidepressant Incomplete and Non-responders With Treatment Resistant Depression (ASCERTAIN-TRD)
Brief Title: Comparative Effectiveness Research Trial for Antidepressant Incomplete and Non-responders With TRD
Acronym: ASCERTAINTRD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, George I. Papakostas, Scientific Director, MGH Clinical Trial Network and Institute (CTNI), Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015P002430
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Treatment Resistant Major Depressive Disorder
MeSH Terms: interventions — Aripiprazole; Transcranial Magnetic Stimulation; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Aripiprazole Augmentation (Experimental): Patients randomized to this treatment arm will be instructed to continue all permitted psychotropics at their current dose throughout the 8-week trial and initiate adjunctive aripiprazole. The starting dose will be 5mg daily. The dose may be reduced to as low as 2mg for tolerability issues (this will be the lowest dose permitted for continuation in the trial). The dose may be adjusted in 2 or 5mg increments. The minimum time per increment will be 7 days. The maximum dose will be set at 15mg daily. For patients who are not on potent cytochrome 2D6 inhibitors (such as paroxetine, fluoxetine, duloxetine) or on potent cytochrome 3A4 inhibitors (such as fluvoxamine and nefazodone) and who are able to tolerate 15mg daily, the maximum dose can be raised to 20mg daily for efficacy.
  Interventions: Drug: Aripiprazole
- rTMS Augmentation (Experimental): Patients randomized to this treatment arm will be instructed to continue all permitted psychotropics at their current dose throughout the 8-week trial. We will use clinical TMS stimulators with focal figure-of-eight coils. We will start by measuring the patient´s motor threshold (MT), which is a measure of cortical excitability used to standardize the intensity of stimulation across subjects.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Switching To Venlafaxine XR (Experimental): Patients randomized to this treatment arm will be instructed to continue all permitted psychotropics throughout the 8-week trial, except for their antidepressant(s). They will be instructed to discontinue all antidepressants and initiate venlafaxine that day, as direct switch to serotonergic antidepressants is well tolerated and avoids loss of precious therapeutic time (Montgomery et al., 2014), including to switching to venlafaxine in STAR*D (Rush et al., 2006b). For patients who do not prefer a direct switch, or when clinically indicated otherwise in the opinion of the site investigator, a gradual tapering during the screening period will be permitted as long as a direct switch to venlafaxine is made on the baseline visit from the final antidepressant dose. The starting dose of venlafaxine will be 75mg daily. The dose may be reduced to as low as 37.5mg for tolerability issues (this will be the lowest dose permitted for continuation in the trial).
  Interventions: Drug: Venlafaxine XR

INTERVENTIONS:
Drug: Aripiprazole — Oral adjunctive therapy with aripiprazole, dose adjusted for effectiveness and tolerability.
  Other Names: Abilify
  Arms: Aripiprazole Augmentation
Device: Repetitive transcranial magnetic stimulation (rTMS) — Adjunctive therapy with transcranial magnetic stimulation, dose adjusted for effectiveness and tolerability.
  Arms: rTMS Augmentation
Drug: Venlafaxine XR — Oral switch therapy with venlafaxine, dose adjusted for effectiveness and tolerability.
  Other Names: Effexor XR
  Arms: Switching To Venlafaxine XR

SUMMARY:
This is a multi-site, randomized, open-label, effectiveness trial comparing three treatment arms for Major Depressive Disorder (MDD) patients with TRD who are currently on ongoing, stable and adequate antidepressant therapy (ADT). Adequate ADT is defined as a therapeutically sufficient dose for a sufficient treatment period, which would be expected to be effective as listed in the MGH Antidepressant Treatment Response Questionnaire (ATRQ). Patients will be randomized in a 1:1:1 fashion to one of three open-label treatment arms: a) aripiprazole augmentation, b) rTMS augmentation, and c) switching to venlafaxine XR or Duloxetine.

ELIGIBILITY:
Inclusion Criteria:

1. women and men ages 18-80,
2. with MDD, of at least 12 weeks duration, according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria confirmed by the Mini International Neuropsychiatric Interview (MINI; Sheehan et al, 1998),
3. have a Montgomery-Asberg Depression Rating Scale (MADRS - Montgomery and Asberg, 1979) score of at least 20 at screen and baseline as assessed by site clinicians,
4. meet criteria for TRD during the current major depressive episode documented in the MGH Antidepressant Treatment History Questionnaire (ATRQ) (Chandler et al., 2010), which will be defined as being non-responders (less than 50% of symptom improvement) to two or more depression treatment trials of adequate dose and duration as defined by the MGH ATRQ,
5. are currently on an antidepressant of adequate dose (as defined by the MGH ATRQ) and duration (at least 8 weeks), with the antidepressant dose being stable over the past four weeks, and with documented (in the MGH ATRQ) non-response (less than 50% improvement) to the current antidepressant.
6. Patients who have passed the MGH CTNI remote assessment, with documentation provided to sites by MGH CTNI.

Exclusion Criteria:

1. pregnant or breastfeeding women, women of childbearing potential who are not using an accepted means of birth control, or women with a positive urine pregnancy test,
2. patients who have received treatment with rTMS, aripiprazole, electroconvulsive therapy (ECT), or venlafaxine during the current episode,
3. patients who express an objection to receiving treatment with at least one of the three treatment arms of our study,
4. patients with any history of bipolar disorder or psychosis (diagnosed by MINI),
5. patients with active alcohol or substance abuse disorders within the past 6 months (diagnosed by MINI),
6. patients with suicidal ideation of the degree that, in the opinion of the evaluating clinician, participation in the study would place them at significantly increased risk of suicide,
7. patients with unstable medical issues of such degree that, in the opinion of the evaluating clinician, participation in the study would place them at significant risk of a serious adverse event, or patients with a screening hemoglobin A1c level greater than 7.5%, or patients with epilepsy, dementia, Parkinson's disease, or Huntington's Disease,
8. patients who have received treatment with vagus nerve stimulation (VNS),
9. patients who have not responded to more than five FDA-approved antidepressant treatment trials of adequate dose and duration during the current episode, or who did not respond to ECT in previous episodes
10. patients on excluded medications,
11. patients with a positive urine screen drug test for a substance for which they do not have a valid prescription for a valid medical reason,
12. patients with currently abnormal thyroid function tests,
13. patients who have received at least one dose of a monoamine oxidase inhibitor (MAOI) four weeks or less prior, and
14. for patients on concomitant psychotropic agents (anticonvulsants, benzodiazepines, hypnotics, opiates, triiodothyronine (T3), modafinil, psychostimulants, buspirone, melatonin, omega-3 fatty acids, folate, l-methylfolate, s-adenosyl methionine, lithium) not on the same dose for at least four weeks prior to study entry or who do not agree to continue at the same dose during the acute phase of the study.
15. Patients who do not meet safety criteria for TMS: history of seizures, cardiac pacemaker, DBS or VNS, brain aneurism clips or other metallic implants in the intracranial space.
16. Also excluded is an individual who has received any administration of ketamine in the current episode for the treatment of depression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 8 weeks
  Assessment of depression severity.

SECONDARY OUTCOMES:
Quality of Life, Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | 8 weeks
  Assessment of quality of life

OTHER OUTCOMES:
Massachusetts General Hospital Cognitive and Physical Symptoms Questionnaire (MGH CPFQ) | 8 weeks
  Assessment of cognitive symptoms

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - The University of Alabama School of Medicine, Birmingham, Alabama
  - Pacific Institute of Medical Research, Los Angeles, California
  - Stanford University, Stanford, California
  - University of South Florida, Tampa, Florida
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - New York University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Roper St. Francis Hospital, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba St. Boniface Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guidetti C, Chaikali S, Trivedi MH, Shelton RC, Iosifescu DV, Thase ME, Jha MK, Mathew SH, DeBattista C, Dokucu ME, Brawman-Mintzer O, Hernandez Ortiz JM, Currier GW, McCall WV, Modirrousta M, Macaluso M, Bystritsky A, Vila-Rodriguez F, Nelson EB, Yeung AS, MacGregor LC, Carmody T, Fava M, Papakostas GI. Comparative Effectiveness Research Trial for Antidepressant Incomplete and Nonresponders With Treatment Resistant Depression (ASCERTAIN-TRD): Effect of Aripiprazole or Repetitive Transcranial Magnetic Stimulation Augmentation Versus Switching to the Antidepressant Venlafaxine on Quality of Life. J Clin Psychiatry. 2025 Aug 11;86(3):24m15614. doi: 10.4088/JCP.24m15614. PMID 40801757
- [Derived] Papakostas GI, Trivedi MH, Shelton RC, Iosifescu DV, Thase ME, Jha MK, Mathew SJ, DeBattista C, Dokucu ME, Brawman-Mintzer O, Currier GW, McCall WV, Modirrousta M, Macaluso M, Bystritsky A, Rodriguez FV, Nelson EB, Yeung AS, Feeney A, MacGregor LC, Carmody T, Fava M. Comparative effectiveness research trial for antidepressant incomplete and non-responders with treatment resistant depression (ASCERTAIN-TRD) a randomized clinical trial. Mol Psychiatry. 2024 Aug;29(8):2287-2295. doi: 10.1038/s41380-024-02468-x. Epub 2024 Mar 7. PMID 38454079